CLINICAL TRIAL: NCT06548048
Title: A Randomized, Double-blind, Parallel Study to Examine the Effects of N-trans-caffeoyl Tyramine and N-trans-feruloyl Tyramine Bioactives on Fat Oxidation in Adult Women With Overweight and Obesity
Brief Title: Dietary Supplementation on Fat Oxidation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brightseed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO-2406
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Treatment (Placebo Comparator)
  Interventions: Dietary Supplement: Microcrystaline cellulose
- Active high dose of plant derived phenolics (Active Comparator)
  Interventions: Dietary Supplement: Dietary supplement containing plant derived phenolics

INTERVENTIONS:
Dietary Supplement: Dietary supplement containing plant derived phenolics — Dietary supplement containing plant derived phenolics
  Arms: Active high dose of plant derived phenolics
Dietary Supplement: Microcrystaline cellulose — Microcrystaline cellulose (MCC)
  Arms: Placebo Treatment

SUMMARY:
The purpose of this pilot study is to evaluate the effects of 4 weeks of daily consumption of encapsulated N-trans-caffeoyl tyramine (NCT) and N-trans-feruloyl tyramine (NFT) at a dose of 120 mg/d on measures of fat oxidation in women with overweight or obesity. The hypothesis is that fat oxidation at rest (measured via indirect calorimetry) and over a 24 h period (measured via d31-palmitic acid stable isotope tracer) will be higher in the group receiving the active study product compared to the control product at the end of the 4-week consumption period.

ELIGIBILITY:
Inclusion Criteria

1. Female, ≥18 and <50 years of age at visit 1 (day -28).
2. Body mass index (BMI) of ≥29.0 kg/m2 to <40.0 kg/m2 at visit 1 (day -28).
3. No health conditions that would prevent fulfilling the study requirements as judged by the Investigator on the basis of medical history.
4. History of regular menstrual cycles with menses (21-35 d per cycle) for at least 3 months prior to visit 1 (day -28).
5. Stable use of non-weight loss (e.g., semaglutide) prescription medications allowed, where stable use is defined as the same class of medication and dose for at least 90 d prior to visit 1 (day -28).
6. Willing to discontinue any dietary supplement use (except for conventional once daily vitamin/mineral supplement[s]), for one week prior to visit 2 and throughout the study.
7. Non-user or former user (cessation ≥12 months) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) with no plans to begin use during the study period.
8. Willing to maintain habitual diet (with the exception of restricted foods/beverages) throughout the study period.
9. Willing to use personal web-based device (e.g., smart phone, tablet, or laptop) with operating system (Android version 12.0 or newer; iOS version 16 or newer) capable of downloading the Cronometer app for diet records.
10. Willing to adhere to all study procedures and signs forms providing informed consent to participate in the study and authorization to release relevant protected health information to the Clinical Investigator.

Exclusion Criteria

1. Unwilling to wear a tampon during the collection of the 24-h urine samples when these collections occur during the time of menstruation
2. Weight loss or gain ≥4.5 kg within 90 days of visit 1 (day -28).
3. Use of weight loss medications within 90 days of visit 1 (day -28).
4. Any health condition that would prevent the participant from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history. Health conditions may include history or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
5. History of gastrointestinal surgery (e.g., bariatric surgery) or cosmetic procedures (e.g., liposuction) for weight/fat reducing purposes.
6. Use of dietary supplements or related products that, in the judgment of the Investigator, are likely to markedly affect weight loss or appetite within 30 days of visit 1.
7. History of extreme dietary habits (e.g., Atkins diet, etc.), as judged by the Investigator.
8. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
9. Current medical diagnosis of type 1 or type 2 diabetes mellitus.
10. History of a chronic gastrointestinal disorder, such as peptic ulcer disease or malabsorption syndrome (mild lactose intolerance or gastroesophageal reflux diseases are acceptable).
11. History of liver disease with exception of non-alcoholic fatty livery disease (NAFLD).
12. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at visit 1.
13. Habitual use (i.e., daily) of marijuana and hemp products including CBD products within 30 days of visit 1.
14. History or presence of cancer (including any malignant GI polyps) within 2 years of visit 1, except for non-melanoma skin cancer.
15. Known intolerance or sensitivity to any ingredients in the study products.
16. Exposure to any non-registered drug product within 30 days prior to visit 1.
17. Signs or symptoms of an active infection of clinical relevance* within 5 days of visit 1. The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to visit 1.
18. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source document.
19. Recent history (within 12 months of visit 1) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz. beer, 5 oz. wine, or 1½ oz. distilled spirits).
20. Any condition the Investigator believes would interfere with her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

    * If an infection occurs during the study period, test visits will be rescheduled until signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to the scheduled study visits.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
% deuterium (2H) label from oxidation of d31-palmitic acid | Day 1 and Day 28 (each day measurements are done in multiple timepoints of Hour 0, Hour 3, Hour 4, Hour 8, and Hour 24)
  Percentage recovery of the deuterium (2H) label from oxidation of d31-palmitic acid to water in urine samples collected

SECONDARY OUTCOMES:
Change in indirect calorimetry measures | day 1 and day 28
  Resting metabolic rate (RMR; kcals/d) derived from the Weir equation
Change in indirect calorimetry measures | day 1 and day 28
  Substrate utilization associated with RMR derived from the Respiratory Exchange Ratio (RER)
Change in cardiometabolic parameters | day 1 and day 28
  Fasting free fatty acids
Change in cardiometabolic parameters | day 1 and day 28
  Fasting NMR lipoproteins
Change in cardiometabolic parameters | day 1 and day 28
  Fasting Glucose
Change in cardiometabolic parameters | day 1 and day 28
  Fasting Insuline
Change in body weight | day 1 and day 28
  Change in body weight measured in scale

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No